CLINICAL TRIAL: NCT03155880
Title: National Health and Nutrition Examination Survey (NHANES), Obesity Heterogeneity Study
Brief Title: Obesity Heterogeneity Study
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 000001
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will assess the heterogeneity of obese individuals in the United States to help researchers, clinicians and policymakers to establish goals for obesity treatment and identify whether differing interventions may be needed.

DETAILED DESCRIPTION:
Guidelines for obesity set common targets for interventions and goals around weight loss, and randomized trials and epidemiologic studies of obesity tend to consider obesity to be a homogeneous entity . The investigators will analyze data from the 2011-2012 wave of the NHANES. Obesity will be defined as having a body mass index greater than or equal to 30 Kg/m2. The investigators aim to identify obese sub-groups according to demographic factors, clinical conditions and behavioral characteristics. Results of this type of analysis will shed light on an important gap in the way that obesity interventions and guidelines are developed and will be an important step in beginning the discussion towards this important area.

ELIGIBILITY:
Inclusion Criteria:

* All

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analyses presented in this report included obese adult participants >=20 years of age, giving a sample size of 1,873 (90% of obese participants). Due to missing data in the covariates, the final analytical sample size was 1,685 (90 % of intended sample).
Sampling Method: Probability Sample
Enrollment: 1685 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Obesity | One day. The body measures data were collected, in the Mobile Examination Center (MEC), by trained health technicians.
  : NHANES collects objective physical examination data for each respondent in the sample, in mobile examination centers for standardization purposes. Body Mass Index (BMI) was calculated as weight in kilograms divided by height in meters squared, and then rounded to one decimal place. Participants were classified as obese using World Health Organization cut-offs for BMI (i.e. ≥30 kg/m2).

IPD SHARING:
Plan to Share IPD: No